CLINICAL TRIAL: NCT02879305
Title: A Phase 3 Randomized, Open-label (Sponsor-blind), Active-controlled, Parallel-group, Multi-center, Event Driven Study in Dialysis Subjects With Anemia Associated With Chronic Kidney Disease to Evaluate the Safety and Efficacy of Daprodustat Compared to Recombinant Human Erythropoietin, Following a Switch From Erythropoietin-stimulating Agents
Brief Title: Anemia Studies in Chronic Kidney Disease: Erythropoiesis Via a Novel Prolyl Hydroxylase Inhibitor Daprodustat-Dialysis (ASCEND-D)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200807; 2016-000541-31 (EudraCT Number)
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Anaemia; Aspergillosis, Allergic Bronchopulmonary
Keywords: erythropoiesis stimulating agents; GSK1278863; daprodustat; anemia; chronic kidney disease; hemoglobin; recombinant human erythropoietin
MeSH Terms: conditions — Anemia; Aspergillosis, Allergic Bronchopulmonary; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daprodustat (Experimental): Participants will receive oral daprodustat once daily.
  Interventions: Drug: Daprodustat; Drug: Placebo; Drug: Iron therapy
- rhEPO (Active Comparator): Participants on peritoneal dialysis (PD) will be administered darbepoetin alfa subcutaneously (SC) and participants on hemodialysis (HD) will be administered epoetin alfa intravenously (IV).
  Interventions: Drug: rhEPO; Drug: Placebo; Drug: Iron therapy

INTERVENTIONS:
Drug: Daprodustat — Daprodustat dose is based on prior ESA dose, the dose is adjusted thereafter in order to achieve the target range.
  Arms: Daprodustat
Drug: rhEPO — The initial ESA dose is based on converting the prior ESA dose to the nearest available study rhEPO dose and is administered IV. The dose is adjusted thereafter in order to achieve the target range.
  Arms: rhEPO
Drug: Placebo — Oral placebo tablets will be taken from Week -4 up to randomization (Day 1).
Drug: Iron therapy — Participants will receive supplemental iron therapy if ferritin is <=100 ng/mL or TSAT is <=20%. The investigator will choose the route of administration and dose of iron.

SUMMARY:
The purpose of this multi-center event-driven study in participants with anemia associated with chronic kidney disease (CKD) to evaluate the safety and efficacy of daprodustat.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 99 years of age (inclusive).
* Erythropoietin-stimulating agents (ESAs): Use of any approved ESA for at least the 6 weeks prior to screening and between screening and randomization.
* Hgb concentration: On Week -8: Hgb 8 to 12 grams per deciliter (g/dL). On randomization (Day 1): Hgb 8 to 11 g/dL and receiving at least the minimum ESA dose. Hgb >11 g/dL to 11.5 g/dL and receiving greater than the minimum ESA dose.
* Dialysis: On dialysis >90 days prior to screening and continuing on the same mode of dialysis from screening (Week -8) through to randomization (Day 1).
* Frequency of Dialysis: Hemodialysis (HD) >=2 times/week and peritoneal dialysis (PD) >=5 times/week. Home hemodialysis >=2 times/week.
* Compliance with placebo [randomization (Day 1) only]: >=80% and <=120% compliance with placebo during run-in period.
* Informed consent (screening only): capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Kidney transplant: Planned living-related or living-unrelated kidney transplant within 52 weeks after study start (Day 1).
* Ferritin: <=100 nanograms (ng)/milliliter (mL) (<=100 micrograms/liter [L]) at screening.
* Transferrin saturation (TSAT) (screening only): <=20%.
* Aplasias: History of bone marrow aplasia or pure red cell aplasia.
* Other causes of anemia: Untreated Pernicious anemia, thalassemia major, sickle cell disease or myelodysplastic syndrome.
* Gastrointestinal (GI) bleeding: Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease or clinically significant GI bleeding <=4 weeks prior to screening through to randomization (Day 1).
* MI or acute coronary syndrome: <=4 weeks prior to screening through to randomization (Day 1).
* Stroke or transient ischemic attack: <=4 weeks prior to screening through to randomization (Day 1).
* Heart failure (HF): Chronic Class IV HF, as defined by the New York Heart Association (NYHA) functional classification system.
* Current uncontrolled hypertension: Current uncontrolled hypertension as determined by the investigator that would contraindicate the use of recombinant human erythropoietin (rhEPO).
* Bazett's corrected QT interval (QTcB) (Day 1): QTcB >500 millisecond (msec), or QTcB >530 msec in subjects with bundle branch block. There is no QT Interval Corrected for Heart Rate (QTc) exclusion for subjects with a predominantly ventricular paced rhythm.
* Alanine transaminase (ALT): >2x upper limit of normal (ULN) at screening.
* Bilirubin: >1.5xULN at screening.
* Current unstable liver or biliary disease per investigator assessment, generally defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Malignancy: History of malignancy within the 2 years prior to screening through to randomization (Day 1) or currently receiving treatment for cancer, or complex kidney cyst (example [e.g.] Bosniak Category II F, III or IV) > 3 centimeter (cm); with the exception of localized squamous cell or basal cell carcinoma of the skin that has been definitively treated >=4 weeks prior to screening.
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product, or epoetin alfa or darbepoetin alfa.
* Drugs and supplements: Use of strong inhibitors of Cytochrome P4502C8 (CYP2C8) (e.g., gemfibrozil) or strong inducers of CYP2C8 (e.g., rifampin/rifampicin).
* Other study participation: Use of other investigational agent or device prior to screening through to randomization (Day 1).
* Prior treatment with daprodustat: Any prior treatment with daprodustat for treatment duration of >30 days.
* Females only: Subject is pregnant [as confirmed by a positive serum human chorionic gonadotrophin (hCG) test for females of reproductive potential (FRP) only], subject is breastfeeding, or subject is of reproductive potential and does not agree to follow one of the contraceptive options listed in the List of Highly Effective Methods for Avoiding Pregnancy.
* Other Conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the subject at unacceptable risk, which may affect study compliance (e.g., intolerance to rhEPO) or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2964 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (385):
- United States (106):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Pine Bluff, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, El Centro, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Fairfield, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Granada Hills, California
  - GSK Investigational Site, Hacienda Heights, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, La Palma, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Lynwood, California
  - GSK Investigational Site, Montebello, California
  - GSK Investigational Site, Monterey Park, California
  - GSK Investigational Site, Moreno Valley, California
  - GSK Investigational Site, Norco, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Ontario, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Luis Obispo, California
  - GSK Investigational Site, Santa Clarita, California
  - GSK Investigational Site, Simi Valley, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Yorba Linda, California
  - GSK Investigational Site, Middlebury, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Gardens, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Spring Hill, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Crystal Lake, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Merrillville, Indiana
  - GSK Investigational Site, Michigan City, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Greenbelt, Maryland
  - GSK Investigational Site, Takoma Park, Maryland
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Pontiac, Michigan
  - GSK Investigational Site, Roseville, Michigan
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, Florissant, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Portsmouth, New Hampshire
  - GSK Investigational Site, Gallup, New Mexico
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Flushing, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Ridgewood, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Yonkers, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Clyde, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Roseburg, Oregon
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Sumter, South Carolina
  - GSK Investigational Site, Cordova, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lufkin, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Bluefield, West Virginia
  - GSK Investigational Site, Shorewood, Wisconsin
- Argentina (10):
  - GSK Investigational Site, Burzaco, Buenos Aires
  - GSK Investigational Site, Ciudad Evita, Buenos Aires
  - GSK Investigational Site, Pergamino, Buenos Aires
  - GSK Investigational Site, Pilar, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Formosa
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Morón
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (16):
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Kingswood, New South Wales
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Birtinya, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, St Albans, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Murdoch
- Austria (3):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Sankt Pölten
  - GSK Investigational Site, Vienna
- Belgium (8):
  - GSK Investigational Site, Baudour
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Ieper
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
- Brazil (10):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Passo Fundo, Rio Grande do Sul
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Joinville, Santa Catarina
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Feira de Santana
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, São Paulo
- Bulgaria (13):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Dobrich
  - GSK Investigational Site, Gabrovo
  - GSK Investigational Site, Lom
  - GSK Investigational Site, Lovech
  - GSK Investigational Site, Montana
  - GSK Investigational Site, Pazardzhik
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Smolyan
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Veliko Tarnovo
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
- Czechia (8):
  - GSK Investigational Site, Beroun
  - GSK Investigational Site, Frýdek-mistek
  - GSK Investigational Site, Ivančice
  - GSK Investigational Site, Jilemnice
  - GSK Investigational Site, Mariánské Lázně
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Sokolov
- Denmark (5):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Holstebro
  - GSK Investigational Site, Kolding
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Svendborg
- Estonia (3):
  - GSK Investigational Site, Pärnu
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (9):
  - GSK Investigational Site, Annonay
  - GSK Investigational Site, Bois-Guillaume
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Mulhouse
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Tours
- Germany (11):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Bad König, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Cloppenburg, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Kaiserslautern, Rhineland-Palatinate
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Dieburg
  - GSK Investigational Site, Freiburg im Breisgau
  - GSK Investigational Site, Minden
- Greece (9):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Arta
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion-Crete
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Komotini
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Thessaloniki
- Hungary (7):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Eger
  - GSK Investigational Site, Esztergom
  - GSK Investigational Site, Kecskemét
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szigetvár
- India (16):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Calicut
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Chennai, Tamil Nadu
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Gūrgaon
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nadiād
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Secunderabad
  - GSK Investigational Site, Trivandrum
- Italy (16):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Reggio Calabria, Calabria
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Piacenza, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Lecco, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Seriate, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Imola
  - GSK Investigational Site, Mestre
- Malaysia (6):
  - GSK Investigational Site, Batu Caves
  - GSK Investigational Site, George Town
  - GSK Investigational Site, Ipoh
  - GSK Investigational Site, Johor Bahru
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuala Pahang
- Mexico (11):
  - GSK Investigational Site, Saltillo, Coahuila
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Querétaro City, Querétaro
  - GSK Investigational Site, Ciudad de México, State of Mexico
  - GSK Investigational Site, Cuautitlán Izcalli, State of Mexico
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, México, D.F.
  - GSK Investigational Site, Zapopan, Jalisco
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Deventer
  - GSK Investigational Site, Rotterdam
- New Zealand (3):
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Hastings
  - GSK Investigational Site, Otahuhu
- Norway (2):
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
- Poland (12):
  - GSK Investigational Site, Biała Podlaska
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Grójec
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Koło
  - GSK Investigational Site, Kołobrzeg
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Olkusz
  - GSK Investigational Site, Pruszków
  - GSK Investigational Site, Tomaszów Mazowiecki
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Żary
- Portugal (9):
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Corroios
  - GSK Investigational Site, Covilha
  - GSK Investigational Site, Forte Da Casa
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Mirandela
  - GSK Investigational Site, Portimão
  - GSK Investigational Site, Vila Franca de Xira
  - GSK Investigational Site, Vila Real (Lordelo)
- Romania (4):
  - GSK Investigational Site, Arad
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Reşiţa
  - GSK Investigational Site, Târgu Jiu
- Russia (11):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Mytischi
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Volzhsky
  - GSK Investigational Site, Yaroslavl
- GSK Investigational Site, Singapore, Singapore
- GSK Investigational Site, Cape Town, South Africa
- South Korea (13):
  - GSK Investigational Site, Anyang-Si, Gyeonggi-do
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Goyang-si
  - GSK Investigational Site, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
  - GSK Investigational Site, Uijeongbu-si
  - GSK Investigational Site, Wŏnju
- Spain (17):
  - GSK Investigational Site, Majadahonda, Madrid
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Aranda de Duero
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Ciudad Real
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Manises (Valencia)
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Mollet del Vallès
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Sabadell
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valladolid
- Sweden (3):
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Taiwan (7):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Keelung
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien
  - GSK Investigational Site, Zhongzheng Dist., Taipei
- Turkey (Türkiye) (6):
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Antalya
  - GSK Investigational Site, Edirne
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Kayseri
- Ukraine (10):
  - GSK Investigational Site, Chernihiv
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kherson
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolaiv
  - GSK Investigational Site, Ternopil
  - GSK Investigational Site, Zaporizhzhia
  - GSK Investigational Site, Zhytomyr
- United Kingdom (13):
  - GSK Investigational Site, Stevenage, Hertfordshire
  - GSK Investigational Site, Preston, Lancashire
  - GSK Investigational Site, Wolverhampton, West Midlands
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Derby
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Fife
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Salford

REFERENCES:
- [Derived] Cunningham JW, Claggett BL, Lopes RD, McMurray JJV, Perkovic V, Carroll K, Hiemstra T, Khavandi K, Lukas MA, Ranganathan P, Shannon J, van Adelsberg J, Singh AK, Solomon SD. Daprodustat and Heart Failure in CKD. J Am Soc Nephrol. 2024 May 1;35(5):607-617. doi: 10.1681/ASN.0000000000000321. Epub 2024 Feb 22. PMID 38383961
- [Derived] Macdougall IC, Meadowcroft AM, Blackorby A, Cizman B, Cobitz AR, Godoy S, Jha V, Johansen KL, McMahon G, Obrador GT, Wong MG, Singh AK. Regional Variation of Erythropoiesis-Stimulating Agent Hyporesponsiveness in the Global Daprodustat Dialysis Study (ASCEND-D). Am J Nephrol. 2023;54(1-2):1-13. doi: 10.1159/000528696. Epub 2023 Feb 7. PMID 36739866
- [Derived] Singh AK, McCausland FR, Claggett BL, Wanner C, Wiecek A, Atkins MB, Carroll K, Perkovic V, McMurray JJV, Wittes J, Snapinn S, Blackorby A, Meadowcroft A, Barker T, DiMino T, Mallett S, Cobitz AR, Solomon SD. Analysis of on-treatment cancer safety events with daprodustat versus conventional erythropoiesis-stimulating agents-post hoc analyses of the ASCEND-ND and ASCEND-D trials. Nephrol Dial Transplant. 2023 Jul 31;38(8):1890-1897. doi: 10.1093/ndt/gfac342. PMID 36565721
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Singh AK, Carroll K, Perkovic V, Solomon S, Jha V, Johansen KL, Lopes RD, Macdougall IC, Obrador GT, Waikar SS, Wanner C, Wheeler DC, Wiecek A, Blackorby A, Cizman B, Cobitz AR, Davies R, Dole J, Kler L, Meadowcroft AM, Zhu X, McMurray JJV; ASCEND-D Study Group. Daprodustat for the Treatment of Anemia in Patients Undergoing Dialysis. N Engl J Med. 2021 Dec 16;385(25):2325-2335. doi: 10.1056/NEJMoa2113379. Epub 2021 Nov 5. PMID 34739194
- [Derived] Singh AK, Blackorby A, Cizman B, Carroll K, Cobitz AR, Davies R, Jha V, Johansen KL, Lopes RD, Kler L, Macdougall IC, McMurray JJV, Meadowcroft AM, Obrador GT, Perkovic V, Solomon S, Wanner C, Waikar SS, Wheeler DC, Wiecek A. Study design and baseline characteristics of patients on dialysis in the ASCEND-D trial. Nephrol Dial Transplant. 2022 Apr 25;37(5):960-972. doi: 10.1093/ndt/gfab065. PMID 33744933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, open-label (sponsor blind), active-controlled, parallel-group, event-driven study conducted at 431 centers in 35 countries. Participants were randomized to receive daprodustat and recombinant human erythropoietin (rhEPO) (epoetin alfa or darbepoetin alfa).
Pre-assignment Details: A total of 2964 participants were randomized in the study.
Groups:
- Daprodustat: Participants received placebo tablets orally once daily in run-in period from Week -4 up to randomization (Day 1) and subsequently received daprodustat tablets at dose levels of 1, 2, 4, 6, 8, 10, 12, 16 and 24 milligrams (mg) orally once daily until the required number of major adverse cardiovascular event (MACE) occurred, at approximately 45.1 months of randomized treatment. Study treatment was dose-titrated to achieve and maintain hemoglobin in the target range (10 to 11 grams per deciliter [g/dL]).
- rhEPO: Participants received placebo tablets orally once daily in run-in period from Week -4 up to randomization (Day 1) and subsequently received treatment with rhEPO. Participants on hemodialysis received epoetin alfa as intravenous (IV) injection once weekly or three-times weekly with total weekly dose levels ranging from 1500 to 60,000 Units. Participants on peritoneal dialysis received subcutaneous (SC) injection of darbepoetin alfa every 1, 2, or 4 weeks with 4-weekly total dose levels ranging from 20 to 400 microgram (mcg). Darbepoetin could be given by IV injection for peritoneal dialysis participants switching to hemodialysis. Study treatment was dose-titrated to achieve and maintain hemoglobin in the target range (10 to 11 g/dL) and administered until the required number of MACE events occurred, at approximately 45.1 months of randomized treatment.
Period: Overall Study
Arm/Group | Daprodustat | rhEPO
Started | 1487 | 1477
Completed | 1370 | 1366
Not Completed | 117 | 111
Not completed — Investigator Site Closed | 55 | 57
Not completed — Withdrawal by Subject | 44 | 42
Not completed — Lost to Follow-up | 17 | 12
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized (Intent-to-treat [ITT]) Population comprised of all randomized participants. Participants were analyzed according to the treatment to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat | rhEPO | Total
Number analyzed (Participants) | 1487 | 1477 | 2964
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (14.29) | 57.3 (14.65) | 57.2 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 636 | 630 | 1266
  Male | 851 | 847 | 1698
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 19 | 32 | 51
  Asian - Central/South Asian Heritage | 36 | 46 | 82
  Asian - East Asian Heritage | 97 | 86 | 183
  Asian - Japanese Heritage | 3 | 3 | 6
  Asian - South East Asian Heritage | 40 | 45 | 85
  Black or African American | 228 | 233 | 461
  Native Hawaiian or Other Pacific Islander | 26 | 25 | 51
  White - Arabic/North African Heritage | 8 | 14 | 22
  White - White/Caucasian/European Heritage | 987 | 968 | 1955
  Mixed Asian Race | 0 | 1 | 1
  Mixed Race | 43 | 24 | 67

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Adjudicated Major Adverse Cardiovascular Event (MACE) During Cardiovascular (CV) Events Follow-up Time Period: Non-inferiority Analysis
Description: Time to MACE defined as the time to first occurrence of Clinical Events Committee (CEC) adjudicated MACE (composite of all-cause mortality, non-fatal myocardial infarction [MI] and non-fatal stroke) was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) plus (+) 1. The incidence rate per 100 person years calculated as (100 multiplied by [*] number of participants with at least 1 event) divided by [/] first event person-years) is presented along with 95 percent (%) confidence interval (CI). First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 11.07 [9.98 to 12.26] | 11.86 [10.72 to 13.09]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Non-Inferiority — Non-inferiority was achieved if the upper limit of the two-sided 95% CI for the hazard ratio was below the pre-specified non-inferiority margin of 1.25; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.81 to 1.07] — Hazard ratio was estimated using a Cox proportional hazard regression model with treatment group, dialysis type and region as covariates

2. Primary Outcome: Mean Change From Baseline in Hemoglobin (Hgb) Levels During Evaluation Period (Week 28 to Week 52)
Description: Blood samples were collected from participants for hemoglobin measurements. Hemoglobin during the evaluation period was defined as the mean of all available post-randomization hemoglobin values (on and off-treatment) during the evaluation period (Week 28 to Week 52). For the primary analysis, missing post-Baseline hemoglobin values were imputed using pre-specified multiple imputation methods. Change from Baseline was defined as post-Baseline value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1) and evaluation period (Week 28 to Week 52)
Population: All Randomized (ITT) Population.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Grams per deciliter | 0.28 (0.022) | 0.10 (0.022)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% CI for the treatment difference was greater than -0.75 g/dL; Least square (LS) mean difference = 0.18, 95% CI 2-sided [0.12 to 0.24] — Analysis of covariance (ANCOVA) model adjusted for treatment, Baseline Hgb, dialysis type and region along with 95% CI for treatment difference (daprodustat-rhEPO)

3. Secondary Outcome: Time to First Occurrence of Adjudicated MACE During CV Events Follow-up Time Period: Superiority Analysis
Description: Time to MACE defined as the time to first occurrence of CEC adjudicated MACE was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariate. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period. This endpoint was adjusted for multiplicity using the Holm-Bonferonni method.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 11.07 [9.98 to 12.26] | 11.86 [10.72 to 13.09]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.156123, Wald test — The p-value was compared against 0.0125 based on the Holm-Bonferonni adjustment; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.81 to 1.07] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to First Occurrence of Adjudicated MACE or Thromboembolic Event During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated MACE or thromboembolic event (vascular access thrombosis, symptomatic deep vein thrombosis or symptomatic pulmonary embolism) was analyzed using a Cox proportional hazards regression model with with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period. This endpoint was adjusted for multiplicity using the Holm-Bonferonni method.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 15.84 [14.48 to 17.30] | 17.85 [16.38 to 19.42]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.023539, Wald test — The p-value was compared against 0.006250 based on the Holm-Bonferonni adjustment; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.78 to 1.00] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to First Occurrence of Adjudicated MACE or Hospitalization for Heart Failure During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated MACE or hospitalization for heart failure was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period. This endpoint was adjusted for multiplicity using the Holm-Bonferonni method.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 12.98 [11.77 to 14.27] | 13.38 [12.15 to 14.70]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.325797, Wald test — The p-value was compared against 0.025000 based on the Holm-Bonferonni adjustment; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.85 to 1.11] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Mean Average Monthly On-treatment IV Iron Dose Per Participant
Description: Average monthly IV iron dose (milligrams) per participant from Day 1 to Week 52 was determined by calculating the total IV iron dose per participant from treatment start date + 1 to the earliest of (Week 52 visit date, first blood (red blood cell [RBC] or whole blood) transfusion date, and treatment stop date + 1 day) which corresponds to the time while the participant was on randomized treatment and before receiving a blood transfusion. This total IV iron dose was divided by (the number of days from treatment start date + 1 to the earliest of (Week 52 visit date, first blood transfusion date (RBC or whole blood), and treatment stop date +1) / 30.4375 days). This endpoint was adjusted for multiplicity using the Holm-Bonferonni method.
Time Frame: Day 1 to Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Milligrams
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1482 | 1472
Milligrams | 90.8 (3.34) | 99.9 (3.35)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.026947, ANCOVA — The p-value was compared against 0.008333 based on the Holm-Bonferonni adjustment; LS mean difference = -9.1, 95% CI 2-sided [-18.4 to 0.2] — Analysis was carried out by using ANCOVA model with terms for treatment, Baseline monthly IV iron dose, dialysis type and region

7. Secondary Outcome: Time to First Occurrence of Adjudicated All-Cause Mortality During Vital Status for Follow-up Time Period
Description: Time to first occurrence of adjudicated all-cause mortality was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the vital status for follow-up time period.
Time Frame: Up to 3.9 person-years for vital status follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 8.32 [7.39 to 9.32] | 8.59 [7.65 to 9.62]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.3281, Wald test; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.82 to 1.13] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time to First Occurrence of Adjudicated CV Mortality During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated CV mortality was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 3.31 [2.74 to 3.97] | 3.46 [2.88 to 4.14]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.3553, Wald test; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.74 to 1.23] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Time to First Occurrence of Adjudicated Myocardial Infarction (MI) (Fatal and Non-Fatal) During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated MI (fatal and non-fatal) was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 3.34 [2.76 to 4.01] | 4.08 [3.43 to 4.83]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0524, Wald test; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.63 to 1.04] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Time to First Occurrence of Adjudicated Stroke (Fatal and Non-Fatal) During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated stroke (fatal and non-fatal) was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 1.23 [0.89 to 1.66] | 1.48 [1.10 to 1.94]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1927, Wald test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.56 to 1.25] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Number of Participants With Adjudicated MACE or Hospitalization for Heart Failure (Recurrent Events Analysis)
Description: Number of participants with adjudicated MACE or hospitalization for heart failure (recurrent events analysis) is presented, categorized by number of occurrences of adjudicated MACE or hospitalization for heart failure per participant.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Participants
  Occurrences per participant: 0 | 1062 | 1044
  Occurrences per participant: 1 | 315 | 300
  Occurrences per participant: 2 | 72 | 88
  Occurrences per participant: 3 | 25 | 22
  Occurrences per participant: 4 | 3 | 11
  Occurrences per participant: 5 | 4 | 4
  Occurrences per participant: 6 | 4 | 3
  Occurrences per participant: 7 | 0 | 2
  Occurrences per participant: 8 | 0 | 1
  Occurrences per participant: 9 | 1 | 1
  Occurrences per participant: 10 | 1 | 1
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0351, Chi-squared; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.80 to 1.01] — Overall HR is presented using Model 1. Model 1 assumed a common treatment effect, regardless of number of events experienced. HR was estimated using a Prentice, Williams and Peterson(PWP) model, with treatment, dialysis type and region as covariates
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.3258, Chi-squared; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.85 to 1.11] — First Event Hazard ratio is presented using Model 2. Model 2 assumed treatment effect differs by number of events experienced. Hazard Ratio (HR) was estimated using a PWP model, with treatment, dialysis type and region as covariates
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0158, Chi-squared; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.58 to 0.98] — Second Event Hazard ratio is presented using Model 2. Model 2 assumed treatment effect differs by number of events experienced. HR was estimated using a PWP model, with treatment, dialysis type and region as covariates
Statistical Analysis 4: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0981, Chi-squared; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.47 to 1.17] — Third Event Hazard ratio is presented using Model 2. Model 2 assumed treatment effect differs by number of events experienced. HR was estimated using a PWP model, with treatment, dialysis type and region as covariates
Statistical Analysis 5: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.3258, Chi-squared; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.85 to 1.11] — First Event Hazard ratio is presented using Model 3. Model 3 assumed treatment effect for first event differs from a common effect for subsequent events. HR was estimated using a PWP model, with treatment, dialysis type and region as covariates
Statistical Analysis 6: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0058, Chi-squared; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.60 to 0.94] — Subsequent Event Hazard ratio is presented using Model 3. Model 3 assumed treatment effect for first event differs from a common effect for subsequent events. HR was estimated using a PWP model, with treatment, dialysis type and region as covariates

12. Secondary Outcome: Time to First Occurrence of Adjudicated CV Mortality or Non-Fatal MI During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated CV mortality or non-fatal MI was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 5.98 [5.18 to 6.86] | 6.79 [5.94 to 7.73]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0872, Wald test; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.06] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Time to First Occurrence of All-Cause Hospitalization During CV Events Follow-up Time Period
Description: All-cause hospitalization events were hospital admissions recorded on the Hospitalization electronic case report form (eCRF) with a hospitalization duration >=24 hours. Time to first occurrence of all-cause hospitalization was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 43.92 [41.18 to 46.81] | 46.03 [43.17 to 49.04]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1540, Wald test; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.87 to 1.04] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Time to First Occurrence of All-Cause Hospital Re-admission Within 30 Days During CV Events Follow-up Time Period
Description: All-cause hospital re-admissions within 30days are defined as hospital admissions recorded on hospitalization eCRF with hospitalization duration of >=24 hours and admission date within 30days following previous discharge date of all-cause hospitalization event, where previous hospitalization was >=24 hours. Time to first occurrence of all-cause hospital re-admission within 30days was analyzed using Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date)+1. Incidence rate per 100person years calculated as(100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 8.86 [7.85 to 9.95] | 9.67 [8.62 to 10.82]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1244, Wald test; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.77 to 1.07] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Time to First Occurrence of Adjudicated MACE or Hospitalization for Heart Failure or Thromboembolic Events During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated MACE or hospitalization for heart failure or thromboembolic events were analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 17.74 [16.28 to 19.30] | 19.50 [17.94 to 21.16]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0540, Wald test; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.81 to 1.02] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Time to First Occurrence of Adjudicated Hospitalization for Heart Failure During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated hospitalization for heart failure was analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 3.30 [2.72 to 3.97] | 3.01 [2.45 to 3.65]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.7658, Wald test; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.84 to 1.45] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Time to First Occurrence of Adjudicated Thromboembolic Events During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated thromboembolic events were analyzed using a Cox proportional hazards regression model with treatment group, dialysis type and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 3.9 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Events per 100 person years | 5.66 [4.87 to 6.54] | 6.75 [5.88 to 7.72]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0425, Wald test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.02] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Change From Baseline in Post-randomization Hemoglobin Levels at Week 52
Description: Blood samples were collected from participants for hemoglobin measurements. Change from Baseline was defined as post-Baseline value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. Analysis was performed using mixed model repeated measures (MMRM) model fitted from Baseline up to Week 52, excluding values collected during the stabilization period, with factors for treatment, time, dialysis type, region, Baseline hemoglobin and Baseline hemoglobin by time and treatment by time interactions.
Time Frame: Baseline (Pre-dose on Day 1) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1358 | 1347
Grams per deciliter | 0.26 (0.032) | 0.14 (0.032)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% CI for the treatment difference was greater than the pre-specified non-inferiority margin of -0.75 g/dL; LS mean difference = 0.12, 95% CI 2-sided [0.03 to 0.21]

19. Secondary Outcome: Number of Hgb Responders in the Hgb Analysis Range (10 to 11.5 Grams/Deciliter) During Evaluation Period (Week 28 to Week 52)
Description: Mean Hgb during the evaluation period was defined as the mean of all evaluable Hgb values during the evaluation period (Week 28 to Week 52) including any evaluable unscheduled Hgb values that were taken during this time period. Hemoglobin responders were defined as participants with a mean Hgb during the evaluation period that falls within the Hgb analysis range of 10-11.5 g/dL.
Time Frame: Week 28 to Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1238 | 1247
Participants | 903 | 866
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0367, Cochran-Mantel-Haenszel; Difference in response rate = 3.5, 95% CI 2-sided [-0.1 to 7.1] — Cochran-Mantel-Haenszel (CMH) test adjusted for dialysis type, and region was used to compare the number of responders between the treatment groups

20. Secondary Outcome: Percentage of Time With Hemoglobin in the Analysis Range (10 to 11.5 Grams/Deciliter) During Evaluation Period (Week 28 to Week 52): Non-inferiority Analysis
Description: Percentage of days for which a participant's Hgb was within the analysis range of 10-11.5 g/dL (both inclusive) during the evaluation period (Week 28 to Week 52), including any unscheduled evaluable Hgb values that were taken during this time period was calculated. Percentage of time in the analysis range during evaluation period is calculated as time in range during the evaluation period / [Earlier of (Date of the last evaluable Hgb value, Week 52 visit date) - Later of (Date of the first evaluable Hgb value that between Week 16 and Week 52 inclusive, Week 28 visit date)].
Time Frame: Week 28 to Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1202 | 1224
Percentage of days | 60.9 [0.0 to 100.0] | 59.4 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% confidence interval for the treatment difference was greater than non-inferiority margin of -15%; Median Difference (Final Values) = 1.06, 95% CI 2-sided [0.00 to 3.86] — Hodges-Lehmann estimate of the treatment difference (daprodustat-rhEPO) and associated two-sided asymptotic 95% CI is presented

21. Secondary Outcome: Percentage of Time With Hemoglobin in the Analysis Range (10 to 11.5 Grams/Deciliter) During Evaluation Period (Week 28 to Week 52): Superiority Analysis
Description: as for outcome 20
Time Frame: Week 28 to Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1202 | 1224
Percentage of days | 60.9 [0.0 to 100.0] | 59.4 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0805, van Elteren test; Probability = 0.52, 95% CI 2-sided [0.49 to 0.54] — Mann-Whitney estimate (Probability) of the treatment effect has been presented

22. Secondary Outcome: Percentage of Time With Hemoglobin in the Analysis Range (10 to 11.5 Grams/Deciliter) During Maintenance Period (Week 28 to End of Study): Non-inferiority Analysis
Description: Percentage of days for which a participant's Hgb was within the analysis range of 10-11.5 g/dL (both inclusive) during the maintenance period (Week 28 to end of study), including any unscheduled evaluable Hgb values that were taken during this time period was calculated. Percentage of time in the analysis range during maintenance period is calculated as time in range during the maintenance period / [Earlier of (Date of the last evaluable Hgb value, End of study date)- Later of (Date of the first evaluable Hgb value that is on or after week 16, Week 28 visit date)].
Time Frame: Week 28 to end of study (3.9 person-years for follow-up time period)
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1203 | 1224
Percentage of days | 60.9 [0.0 to 100.0] | 57.7 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Non-Inferiority — [test comment as in outcome 20, analysis 1]; Median Difference (Final Values) = 2.18, 95% CI 2-sided [0.28 to 4.05] — [estimate comment as in outcome 20, analysis 1]

23. Secondary Outcome: Percentage of Time With Hemoglobin in the Analysis Range (10 to 11.5 Grams/Deciliter) During Maintenance Period (Week 28 to End of Study): Superiority Analysis
Description: as for outcome 22
Time Frame: Week 28 to end of study (3.9 person-years for follow-up time period)
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1203 | 1224
Percentage of days | 60.9 [0.0 to 100.0] | 57.7 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0139, van Elteren test; Probability = 0.53, 95% CI 2-sided [0.50 to 0.55] — Mann-Whitney estimate (Probability) of the treatment effect has been presented

24. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Mean Arterial Blood Pressure (MAP) at Week 52
Description: SBP, DBP and MAP were measured in a semi-supine or seated position in the dialysis chair after at least a 5-minutes of rest. MAP is the average BP in an individual's arteries during a single cardiac cycle. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. Analysis was performed using MMRM model with treatment group + time + dialysis type + region + Baseline value + Baseline value*time + treatment group*time, using an unstructured covariance matrix. Data for post-dialysis BP measurements have been presented.
Time Frame: Baseline (Week -4) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1455 | 1442
Millimeter of mercury
  SBP | -0.61 (0.582) | -0.93 (0.578)
  DBP | -1.04 (0.326) | -0.58 (0.324)
  MAP | -0.89 (0.370) | -0.71 (0.368)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.6551, MMRM; LS mean difference = 0.33, 95% CI 2-sided [-1.28 to 1.94] — The difference in change from Baseline in SBP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in means between arms
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1586, MMRM; LS mean difference = -0.46, 95% CI 2-sided [-1.36 to 0.44] — The difference in change from Baseline in DBP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in means between arms
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.3646, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-1.20 to 0.84] — The difference in change from Baseline in MAP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in means between arms

25. Secondary Outcome: Change From Baseline in SBP, DBP, MAP at End of Treatment
Description: SBP, DBP and MAP were measured in a semi-supine or seated position in the dialysis chair after at least a 5-minutes of rest. MAP is an average BP in an individual's arteries during a single cardiac cycle. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. This analysis was carried out by using ANCOVA model with terms for treatment group, dialysis type, region and Baseline value. Data for post-dialysis BP measurements have been presented.
Time Frame: Baseline (Week -4) and 45.1 months
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1468 | 1454
Millimeter of mercury
  SBP | -0.43 (0.554) | -0.43 (0.557)
  DBP | -0.92 (0.310) | -1.37 (0.312)
  MAP | -0.75 (0.350) | -1.06 (0.351)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.5012, ANCOVA; LS mean difference = 0.00, 95% CI 2-sided [-1.54 to 1.54] — For SBP: Treatment group comparisons were based on an ANCOVA model with terms for treatment group, dialysis type, region and Baseline value
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.8451, ANCOVA; LS mean difference = 0.45, 95% CI 2-sided [-0.42 to 1.31] — For DBP: Treatment group comparisons were based on an ANCOVA model with terms for treatment group, dialysis type, region and Baseline value
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.7312, ANCOVA; LS mean difference = 0.31, 95% CI 2-sided [-0.67 to 1.28] — For MAP: Treatment group comparisons were based on an ANCOVA model with terms for treatment group, dialysis type, region and Baseline value

26. Secondary Outcome: Blood Pressure (BP) Exacerbation Event Rate Per 100 Participant Years
Description: BP exacerbation was defined (based on post-dialysis) as: SBP >= 25 millimeter of mercury (mmHg) increased from Baseline or SBP >=180 mmHg; DBP >=15 mmHg increased from Baseline or DBP >=110 mmHg. The BP exacerbation events per 100 participant years was estimated using the negative binomial model with treatment, dialysis type and region as covariates and the logarithm of time on-treatment as an offset variable. Data for post-dialysis BP measurements have been presented.
Time Frame: Day 1 to end of study (3.9 person-years for follow-up time period)
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant years
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1470 | 1458
Events per 100 participant years | 207.13 [188.83 to 227.21] | 206.38 [187.88 to 226.71]
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.5290, Negative binomial model; Ratio of exacerbation rate = 1.00, 95% CI 2-sided [0.91 to 1.11] — Ratio of model estimated exacerbation rates and CIs were estimated using a negative binomial model for the treatment group comparison

27. Secondary Outcome: Number of Participants With at Least One BP Exacerbation Event During Study
Description: BP exacerbation was defined as: SBP >= 25 mmHg increased from Baseline or SBP >=180 mmHg; DBP >=15 mmHg increased from Baseline or DBP >=110 mmHg. Number of participants with at least one BP exacerbation event is presented.
Time Frame: Day 1 to end of study (3.9 person-years for follow-up time period)
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1480 | 1470
Participants | 1191 | 1186

28. Secondary Outcome: Percentage of Participants Permanently Stopping Randomized Treatment Due to Meeting Rescue Criteria
Description: Percentage of participants permanently stopping randomized treatment due to meeting rescue criteria has been presented.
Time Frame: Day 1 to 45.1 months
Population: All Randomized (ITT) Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1487 | 1477
Percentage of participants | 3.6 | 3.6
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.5772, Wald test; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.71 to 1.52] — Hazard ratio was estimated using a Cox proportional hazard regression model adjusted for treatment group, dialysis type and region

29. Secondary Outcome: Change From Baseline in On-Treatment Physical Component Score (PCS) Using Short Form (SF)-36 Health-related Quality of Life (HRQoL) Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). The PCS is an average score derived from 4 domains (physical functioning, role-physical, bodily pain and general health) representing overall physical health. PCS ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 990 | 943
Scores on a scale
  Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Week 8, n=982,936 | 0.30 (0.205) | 0.01 (0.210)
  Week 12, n=990,943 | 0.33 (0.203) | -0.27 (0.207)
  Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Week 28, n=836,819 | -0.23 (0.229) | -0.57 (0.232)
  Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Week 52, n=729,707 | -0.52 (0.248) | -1.05 (0.252)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1620, MMRM; LS mean difference = 0.29, 95% CI 2-sided [-0.29 to 0.86] — Week 8: Model was fitted from Baseline up to Week 52 and the model adjusted Week 8 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0180, MMRM; LS mean difference = 0.61, 95% CI 2-sided [0.04 to 1.18] — Week 12: Model was fitted from Baseline up to Week 52 and the model adjusted Week 12 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1530, MMRM; LS mean difference = 0.33, 95% CI 2-sided [-0.31 to 0.97] — Week 28: Model was fitted from Baseline up to Week 52 and the model adjusted Week 28 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0686, MMRM; LS mean difference = 0.53, 95% CI 2-sided [-0.17 to 1.22] — Week 52: Model was fitted from Baseline up to Week 52 and the model adjusted Week 52 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions

30. Secondary Outcome: Change From Baseline in On-Treatment Mental Component Score (MCS) Using SF-36 HRQoL Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). MCS is an average score derived from 4 domains (vitality, social functioning, role-emotional and mental health) representing overall mental health. MCS ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 990 | 943
Scores on a scale
  Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Week 8, n=982,936 | -0.38 (0.254) | -0.21 (0.260)
  Week 12, n=990,943 | -0.55 (0.262) | -0.72 (0.268)
  Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Week 28, n=836,819 | -1.25 (0.286) | -1.23 (0.290)
  Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Week 52, n=729,707 | -1.63 (0.311) | -1.03 (0.316)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.6807, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.88 to 0.54] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.3256, MMRM; LS mean difference = 0.17, 95% CI 2-sided [-0.57 to 0.91] — [estimate comment as in outcome 29, analysis 2]
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.5144, MMRM; LS mean difference = -0.01, 95% CI 2-sided [-0.81 to 0.78] — [estimate comment as in outcome 29, analysis 3]
Statistical Analysis 4: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.9120, MMRM; LS mean difference = -0.60, 95% CI 2-sided [-1.47 to 0.27] — [estimate comment as in outcome 29, analysis 4]

31. Secondary Outcome: Change From Baseline in On-Treatment SF-36 HRQoL Scores for Bodily Pain, General Health, Mental Health, Role-Emotional, Role-Physical, Social Functioning at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: bodily pain, general health, mental health, role-emotional (role limitations caused by emotional problems), role-physical (role limitations caused by physical problems), social functioning (Social fun), physical functioning (Phy. fun) and vitality. Each domain is scored from 0 (poorer health) to 100 (better health). Each domain score ranges from 0 to 100, higher score indicates a better health state and better functioning. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 990 | 943
Scores on a scale
  Bodily pain: Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Bodily pain: Week 8, n=982,936 | -0.13 (0.265) | 0.12 (0.272)
  Bodily pain: Week 12, n=990,943 | 0.20 (0.267) | -0.39 (0.274)
  Bodily pain: Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Bodily pain: Week 28, n=836,819 | -0.70 (0.297) | -0.74 (0.301)
  Bodily pain: Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Bodily pain: Week 52, n=729,707 | -1.12 (0.313) | -1.39 (0.318)
  General health: Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  General health: Week 8, n=982,936 | -0.39 (0.208) | -0.65 (0.213)
  General health: Week 12, n=990,943 | -0.59 (0.210) | -1.04 (0.215)
  General health: Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  General health: Week 28, n=836,819 | -1.32 (0.232) | -0.99 (0.235)
  General health: Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  General health: Week 52, n=729,707 | -1.51 (0.251) | -1.22 (0.255)
  Mental health: Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Mental health: Week 8, n=982,936 | -0.43 (0.238) | -0.47 (0.244)
  Mental health: Week 12, n=990,943 | -0.86 (0.247) | -0.81 (0.253)
  Mental health: Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Mental health: Week 28, n=836,819 | -1.30 (0.267) | -1.43 (0.270)
  Mental health: Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Mental health: Week 52, n=729,707 | -1.97 (0.296) | -1.16 (0.301)
  Role-emotional: Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Role-emotional: Week 8, n=982,936 | -0.10 (0.310) | -0.02 (0.317)
  Role-emotional: Week 12, n=990,943 | -0.17 (0.311) | -0.53 (0.318)
  Role-emotional: Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Role-emotional: Week 28, n=836,819 | -0.95 (0.335) | -0.90 (0.339)
  Role-emotional: Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Role-emotional: Week 52, n=729,707 | -0.83 (0.358) | -0.92 (0.363)
  Role-physical: Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Role-physical: Week 8, n=982,936 | 0.40 (0.241) | 0.32 (0.246)
  Role-physical: Week 12, n=990,943 | 0.48 (0.239) | 0.08 (0.245)
  Role-physical: Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Role-physical: Week 28, n=836,819 | -0.10 (0.257) | -0.39 (0.260)
  Role-physical: Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Role-physical: Week 52, n=729,707 | -0.21 (0.285) | -0.60 (0.289)
  Social functioning: Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Social functioning: Week 8, n=982,936 | 0.24 (0.241) | 0.38 (0.247)
  Social functioning: Week 12, n=990,943 | 0.25 (0.255) | -0.44 (0.261)
  Social functioning: Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Social functioning: Week 28, n=836,819 | -0.61 (0.280) | -0.94 (0.283)
  Social functioning: Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Social functioning: Week 52, n=729,707 | -1.12 (0.315) | -1.14 (0.320)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.7432, MMRM; LS mean difference = -0.25, 95% CI 2-sided [-0.99 to 0.50] — Bodily pain,Week8: Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0631, MMRM; LS mean difference = 0.58, 95% CI 2-sided [-0.16 to 1.33] — Bodily pain,Week12: Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.4604, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-0.79 to 0.87] — Bodily pain,Week28: Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.2688, MMRM; LS mean difference = 0.28, 95% CI 2-sided [-0.60 to 1.15] — Bodily pain,Week52: Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 5: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1918, MMRM; LS mean difference = 0.26, 95% CI 2-sided [-0.32 to 0.84] — General health,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 6: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0677, MMRM; LS mean difference = 0.45, 95% CI 2-sided [-0.14 to 1.04] — General health,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 7: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.8386, MMRM; LS mean difference = -0.33, 95% CI 2-sided [-0.98 to 0.32] — General health,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 8: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.7928, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.99 to 0.41] — General health,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 9: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.4537, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-0.63 to 0.71] — Mental health,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 10: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.5548, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.74 to 0.65] — Mental health,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 11: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.3626, MMRM; LS mean difference = 0.13, 95% CI 2-sided [-0.61 to 0.88] — Mental health,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 12: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.9721, MMRM; LS mean difference = -0.81, 95% CI 2-sided [-1.64 to 0.02] — Mental health,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 13: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.5789, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.96 to 0.78] — Role-emotional,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 14: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.2054, MMRM; LS mean difference = 0.37, 95% CI 2-sided [-0.51 to 1.24] — Role-emotional,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 15: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.5389, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.98 to 0.89] — Role-emotional,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 16: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.4289, MMRM; LS mean difference = 0.09, 95% CI 2-sided [-0.91 to 1.09] — Role-emotional,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 17: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.4096, MMRM; LS mean difference = 0.08, 95% CI 2-sided [-0.60 to 0.75] — Role-physical,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 18: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1196, MMRM; LS mean difference = 0.40, 95% CI 2-sided [-0.27 to 1.07] — Role-physical,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 19: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.2093, MMRM; LS mean difference = 0.30, 95% CI 2-sided [-0.42 to 1.01] — Role-physical,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 20: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1674, MMRM; LS mean difference = 0.39, 95% CI 2-sided [-0.40 to 1.19] — Role-physical,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, dialysis type, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 21: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.6585, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.82 to 0.54] — Social fun, Week 8: Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 22: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0293, MMRM; LS mean difference = 0.69, 95% CI 2-sided [-0.03 to 1.40] — Social fun, Week 12: Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 23: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.2057, MMRM; LS mean difference = 0.33, 95% CI 2-sided [-0.45 to 1.11] — Social fun, Week 28: Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 24: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.4849, MMRM; LS mean difference = 0.02, 95% CI 2-sided [-0.86 to 0.90] — Social fun, Week 52: Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions

32. Secondary Outcome: Change From Baseline in On-Treatment Vitality Scores Using SF-36 HRQoL Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). Vitality score ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 990 | 943
Scores on a scale
  Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Week 8, n=982,936 | -0.23 (0.219) | -0.26 (0.224)
  Week 12, n=990,943 | -0.17 (0.227) | -0.51 (0.232)
  Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Week 28, n=836,819 | -0.79 (0.242) | -1.03 (0.245)
  Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Week 52, n=729,707 | -1.19 (0.268) | -1.04 (0.272)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.4621, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.58 to 0.64] — Week 8: Model was fitted from Baseline up to Week 52 and model adjusted Week 8 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1439, MMRM; LS mean difference = 0.35, 95% CI 2-sided [-0.29 to 0.98] — Week 12: Model was fitted from Baseline up to Week 52 and model adjusted Week 12 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.2392, MMRM; LS mean difference = 0.24, 95% CI 2-sided [-0.43 to 0.92] — Week 28: Model was fitted from Baseline up to Week 52 and model adjusted Week 28 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.6545, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.90 to 0.60] — Week 52: Model was fitted from Baseline up to Week 52 and model adjusted Week 52 data has been presented, with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions

33. Secondary Outcome: Change From Baseline in On-Treatment Physical Functioning Domain Scores Using SF-36 HRQoL Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). Physical functioning score ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as on-treatment visit value minus (-) Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 990 | 943
Scores on a scale
  Week 8, n=982,936: number analyzed (Participants) | 982 | 936
  Week 8, n=982,936 | 0.48 (0.237) | -0.16 (0.243)
  Week 12, n=990,943 | 0.11 (0.240) | -0.45 (0.246)
  Week 28, n=836,819: number analyzed (Participants) | 836 | 819
  Week 28, n=836,819 | -0.20 (0.273) | -0.97 (0.277)
  Week 52, n=729,707: number analyzed (Participants) | 729 | 707
  Week 52, n=729,707 | -0.61 (0.291) | -1.19 (0.296)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0290, MMRM; LS mean difference = 0.64, 95% CI 2-sided [-0.02 to 1.31] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0509, MMRM; LS mean difference = 0.56, 95% CI 2-sided [-0.11 to 1.24] — [estimate comment as in outcome 32, analysis 2]
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0237, MMRM; LS mean difference = 0.77, 95% CI 2-sided [0.01 to 1.53] — [estimate comment as in outcome 32, analysis 3]
Statistical Analysis 4: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0828, MMRM; LS mean difference = 0.58, 95% CI 2-sided [-0.24 to 1.39] — [estimate comment as in outcome 32, analysis 4]

34. Secondary Outcome: Change From Baseline in On-Treatment Health Utility EuroQol 5 Dimensions 5 Level (EQ-5D-5L) Questionnaire Score at Week 52
Description: EQ-5D-5L is self-assessment questionnaire,consisting of 5 items covering 5 dimensions (mobility,self care,usual activities,pain/discomfort and anxiety/depression). Each dimension is measured by 5-point Likert scale (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems). Responses for 5 dimensions together formed a 5-figure description of health state (e.g.11111 indicates no problems in all 5 dimensions). Each of these 5 figure health states were converted to a single index score by applying country-specific value set formula that attaches weights to dimensions and levels. Range for EQ-5D-5L index score is -0.594 (worst health) to 1 (full health state). Change from Baseline was calculated as on-treatment visit value-Baseline value. Baseline was latest non-missing pre-dose assessment on or before randomization date.
Time Frame: Baseline (Pre-dose on Day 1) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 333 | 329
Scores on a scale | -0.0198 (0.01179) | -0.0201 (0.01187)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.4939, MMRM; LS mean difference = 0.0003, 95% CI 2-sided [-0.0326 to 0.0331] — MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, region, Baseline value and Baseline value by time and treatment by time interactions

35. Secondary Outcome: Change From Baseline in On-Treatment EuroQol Visual Analogue Scale (EQ-VAS) at Week 52
Description: The EQ VAS records the respondent's self-rated health on a vertical VAS, ranging from 0 to 100, where 0 represents the worst health one can imagine and 100 represents the best health one can imagine. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 333 | 329
Scores on a scale | -1.0 (0.86) | 0.8 (0.87)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.9292, MMRM; LS mean difference = -1.8, 95% CI 2-sided [-4.2 to 0.6] — [estimate comment as in outcome 34, analysis 1]

36. Secondary Outcome: Change From Baseline in On-Treatment Patient Global Impression of Severity (PGI-S) at Weeks 8, 12, 28, 52
Description: The PGI-S is a 1-item questionnaire designed to assess participant's impression of disease severity on a 5-point disease severity scale (0=absent, 1=mild, 2=moderate, 3=severe, or 4=very severe). A higher score indicated worse outcome. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | rhEPO
Number analyzed (Participants) | 1102 | 1073
Scores on a scale
  Week 8, n=1102,1064: number analyzed (Participants) | 1102 | 1064
  Week 8, n=1102,1064 | -0.03 (0.024) | 0.02 (0.025)
  Week 12, n=1102,1073 | 0.02 (0.025) | 0.06 (0.025)
  Week 28, n=934,933: number analyzed (Participants) | 934 | 933
  Week 28, n=934,933 | 0.04 (0.027) | 0.08 (0.027)
  Week 52, n=826,814: number analyzed (Participants) | 826 | 814
  Week 52, n=826,814 | 0.06 (0.029) | 0.11 (0.030)
Statistical Analysis 1: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.0428, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.13 to 0.01] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1155, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.11 to 0.03] — [estimate comment as in outcome 32, analysis 2]
Statistical Analysis 3: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1426, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.12 to 0.03] — [estimate comment as in outcome 32, analysis 3]
Statistical Analysis 4: Comparison: Daprodustat vs rhEPO; Test type: Superiority; p = 0.1152, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.13 to 0.03] — [estimate comment as in outcome 32, analysis 4]

ADVERSE EVENTS:
Time Frame: All-cause mortality, treatment emergent serious adverse events (TESAEs) and non-serious treatment emergent adverse events (TEAEs) were collected up to 3.9 person-years for CV follow-up time period
Description: All-cause mortality used All Randomized (ITT) Population consisting of all randomized participants and analyzed based on treatment to which they were randomized. TESAEs and non-serious TEAEs used Safety Population, which included all randomized participants who received at least 1 dose of treatment and analyzed based on treatment received. Eight participants in All Randomized (ITT) Population did not receive treatment and were excluded from Safety Population.
Arm/Group | Daprodustat | rhEPO
All-Cause Mortality (participants affected / at risk) | 294/1487 | 300/1477
Serious Adverse Events (participants affected / at risk) | 773/1482 | 748/1474
Other Adverse Events (participants affected / at risk) | 830/1482 | 827/1474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=1482) | rhEPO (N=1474)
Pneumonia (Infections and infestations) | 86 (97) | 81 (96)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 36 (43) | 57 (74)
Fluid overload (Metabolism and nutrition disorders) | 42 (53) | 45 (57)
Anaemia (Blood and lymphatic system disorders) | 26 (29) | 41 (52)
Sepsis (Infections and infestations) | 29 (31) | 37 (37)
Acute myocardial infarction (Cardiac disorders) | 30 (33) | 31 (40)
Atrial fibrillation (Cardiac disorders) | 23 (26) | 35 (44)
Hyperkalaemia (Metabolism and nutrition disorders) | 19 (23) | 36 (41)
Peritonitis (Infections and infestations) | 31 (42) | 24 (34)
COVID-19 (Infections and infestations) | 22 (22) | 22 (22)
Cellulitis (Infections and infestations) | 16 (18) | 21 (26)
Cardiac arrest (Cardiac disorders) | 20 (20) | 15 (15)
Angina pectoris (Cardiac disorders) | 18 (19) | 16 (18)
Gangrene (Infections and infestations) | 15 (19) | 19 (28)
Cardiac failure (Cardiac disorders) | 18 (23) | 15 (15)
Cardiac failure congestive (Cardiac disorders) | 18 (19) | 15 (19)
Myocardial infarction (Cardiac disorders) | 11 (11) | 17 (17)
Osteomyelitis (Infections and infestations) | 15 (18) | 13 (16)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 13 (14)
Angina unstable (Cardiac disorders) | 14 (14) | 13 (15)
Hypertension (Vascular disorders) | 16 (18) | 11 (14)
Coronary artery disease (Cardiac disorders) | 10 (11) | 16 (16)
Non-cardiac chest pain (General disorders) | 10 (11) | 16 (23)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 15 (17)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 15 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 12 (12)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 12 (12) | 12 (12)
Hypotension (Vascular disorders) | 5 (5) | 19 (19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 11 (11)
Septic shock (Infections and infestations) | 8 (9) | 16 (17)
Urinary tract infection (Infections and infestations) | 13 (14) | 11 (16)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (13) | 11 (12)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 7 (9) | 15 (25)
Device related infection (Infections and infestations) | 13 (14) | 9 (10)
Gastroenteritis (Infections and infestations) | 9 (9) | 13 (15)
Ischaemic stroke (Nervous system disorders) | 11 (11) | 11 (11)
Fall (Injury, poisoning and procedural complications) | 14 (15) | 7 (7)
Cerebrovascular accident (Nervous system disorders) | 9 (11) | 11 (13)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (10)
Hypoglycaemia (Metabolism and nutrition disorders) | 11 (12) | 9 (10)
Lower respiratory tract infection (Infections and infestations) | 9 (10) | 11 (11)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10)
Staphylococcal sepsis (Infections and infestations) | 10 (10) | 10 (10)
Influenza (Infections and infestations) | 8 (8) | 11 (11)
Peripheral ischaemia (Vascular disorders) | 12 (14) | 7 (7)
Arteriovenous fistula site infection (Infections and infestations) | 12 (13) | 6 (6)
Device malfunction (Product Issues) | 7 (8) | 11 (11)
Syncope (Nervous system disorders) | 5 (6) | 13 (13)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 9 (10) | 8 (10)
Transient ischaemic attack (Nervous system disorders) | 7 (7) | 10 (12)
Bronchitis (Infections and infestations) | 8 (8) | 7 (8)
Pyrexia (General disorders) | 7 (7) | 8 (8)
Staphylococcal bacteraemia (Infections and infestations) | 8 (9) | 7 (9)
Hypertensive urgency (Vascular disorders) | 6 (7) | 8 (10)
Peritonitis bacterial (Infections and infestations) | 6 (6) | 8 (14)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 10 (10)
Cardio-respiratory arrest (Cardiac disorders) | 8 (8) | 5 (5)
Device related sepsis (Infections and infestations) | 7 (11) | 6 (7)
Diabetic foot infection (Infections and infestations) | 7 (7) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 7 (7)
Femur fracture (Injury, poisoning and procedural complications) | 8 (9) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9)
Metabolic encephalopathy (Nervous system disorders) | 3 (3) | 9 (10)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 8 (9)
Urosepsis (Infections and infestations) | 7 (7) | 5 (5)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 7 (9) | 5 (7)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 6 (6) | 5 (7)
Asthenia (General disorders) | 5 (5) | 6 (6)
Bacteraemia (Infections and infestations) | 4 (4) | 7 (7)
Death (General disorders) | 9 (9) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (3)
Dialysis hypotension (Vascular disorders) | 6 (6) | 5 (5)
Hypertensive emergency (Vascular disorders) | 3 (3) | 8 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Staphylococcal infection (Infections and infestations) | 8 (9) | 3 (3)
Vascular access malfunction (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 5 (6) | 5 (5)
Bradycardia (Cardiac disorders) | 2 (2) | 8 (8)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 7 (7)
Extremity necrosis (Vascular disorders) | 3 (4) | 7 (9)
Haematoma (Vascular disorders) | 5 (5) | 5 (6)
Postoperative wound infection (Infections and infestations) | 6 (8) | 4 (4)
Acute left ventricular failure (Cardiac disorders) | 4 (4) | 5 (6)
Aortic stenosis (Vascular disorders) | 2 (2) | 7 (9)
Arteriovenous graft site infection (Infections and infestations) | 4 (4) | 5 (5)
Atrial flutter (Cardiac disorders) | 4 (4) | 5 (5)
Cardiac failure acute (Cardiac disorders) | 8 (8) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 5 (5) | 4 (4)
Endocarditis (Infections and infestations) | 6 (6) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 6 (6)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Hypertensive crisis (Vascular disorders) | 5 (5) | 4 (5)
Seizure (Nervous system disorders) | 4 (4) | 5 (5)
Ascites (Gastrointestinal disorders) | 4 (4) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gastritis erosive (Gastrointestinal disorders) | 7 (7) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 5 (8) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 5 (5) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 6 (6)
Pelvic fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2)
Abscess limb (Infections and infestations) | 4 (4) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 5 (5)
Arteriovenous fistula site pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Blood loss anaemia (Blood and lymphatic system disorders) | 4 (5) | 3 (3)
Cataract (Eye disorders) | 2 (3) | 5 (6)
Catheter site infection (Infections and infestations) | 5 (8) | 2 (2)
Chest pain (General disorders) | 2 (2) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 5 (5)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Fibula fracture (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 4 (5) | 3 (3)
Localised infection (Infections and infestations) | 2 (3) | 5 (5)
Pericardial effusion (Cardiac disorders) | 3 (3) | 4 (6)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Accelerated hypertension (Vascular disorders) | 1 (1) | 5 (6)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 4 (8) | 2 (4)
Arthritis bacterial (Infections and infestations) | 3 (3) | 3 (4)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 4 (4)
Azotaemia (Renal and urinary disorders) | 2 (2) | 4 (4)
Colitis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Encephalopathy (Nervous system disorders) | 2 (2) | 4 (5)
End stage renal disease (Renal and urinary disorders) | 5 (5) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (5) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 5 (5)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Mitral valve incompetence (Cardiac disorders) | 4 (4) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 4 (4) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Post procedural infection (Infections and infestations) | 1 (1) | 5 (5)
Prostatitis (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Thrombosis in device (Product Issues) | 2 (2) | 4 (4)
Vascular device infection (Infections and infestations) | 2 (2) | 4 (5)
Brachiocephalic vein stenosis (Vascular disorders) | 3 (4) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Cerebral infarction (Nervous system disorders) | 2 (2) | 3 (3)
Cholecystitis chronic (Hepatobiliary disorders) | 3 (3) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Diverticulitis (Infections and infestations) | 1 (1) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (1) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 4 (4) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (4) | 2 (2)
Hypertensive encephalopathy (Nervous system disorders) | 3 (3) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Infected skin ulcer (Infections and infestations) | 2 (2) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Intervertebral discitis (Infections and infestations) | 3 (3) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 1 (2) | 4 (4)
Pericarditis (Cardiac disorders) | 2 (2) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 4 (4) | 1 (1)
Pneumonia viral (Infections and infestations) | 2 (2) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (5) | 2 (2)
Subclavian vein stenosis (Vascular disorders) | 3 (7) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Vascular access site infection (Infections and infestations) | 4 (4) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 3 (4)
Anal abscess (Infections and infestations) | 2 (2) | 2 (2)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 2 (4) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Congestive cardiomyopathy (Cardiac disorders) | 3 (3) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 3 (3)
Diabetic gangrene (Infections and infestations) | 2 (3) | 2 (2)
Diabetic gastroparesis (Gastrointestinal disorders) | 3 (4) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dry gangrene (Vascular disorders) | 3 (3) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Escherichia sepsis (Infections and infestations) | 2 (2) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fungal peritonitis (Infections and infestations) | 4 (4) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 2 (2) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 3 (3) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Mental status changes (Psychiatric disorders) | 1 (1) | 3 (3)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 2 (2)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Right ventricular failure (Cardiac disorders) | 2 (2) | 2 (2)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (2) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Sudden cardiac death (General disorders) | 3 (3) | 1 (1)
Sudden death (General disorders) | 3 (3) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
Suspected COVID-19 (Infections and infestations) | 3 (4) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Transaminases increased (Investigations) | 0 (0) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 2 (3) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Device related bacteraemia (Infections and infestations) | 2 (3) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dialysis related complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4)
Ejection fraction decreased (Investigations) | 2 (2) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 2 (2) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 2 (2)
Erysipelas (Infections and infestations) | 2 (2) | 1 (1)
Escherichia infection (Infections and infestations) | 2 (2) | 1 (1)
Facial paralysis (Nervous system disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Haemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Hepatitis C (Infections and infestations) | 0 (0) | 3 (3)
Hungry bone syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 3 (3) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 2 (2)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Klebsiella infection (Infections and infestations) | 2 (2) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 2 (2) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 3 (3) | 0 (0)
Shunt blood flow excessive (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 3 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Steal syndrome (Vascular disorders) | 1 (1) | 2 (2)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 3 (3)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 2 (2)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Troponin increased (Investigations) | 1 (1) | 2 (2)
Vascular access steal syndrome (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal adhesions (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 1 (1)
Acute hepatitis B (Infections and infestations) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis perforated (Infections and infestations) | 2 (2) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 2 (2)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 2 (2)
Atypical pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 2 (4)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Calciphylaxis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Carbuncle (Infections and infestations) | 2 (2) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 2 (3)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cholecystitis infective (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colonic abscess (Infections and infestations) | 1 (1) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Device related thrombosis (General disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 2 (3)
Endometriosis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Gas gangrene (Infections and infestations) | 1 (1) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 2 (4)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic cyst infection (Infections and infestations) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 2 (3) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hyperparathyroidism tertiary (Endocrine disorders) | 2 (4) | 0 (0)
Hypocalcaemic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lung abscess (Infections and infestations) | 0 (0) | 2 (2)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Nervous system disorder (Nervous system disorders) | 2 (2) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (4) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 1 (1)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 0 (0)
Pericarditis uraemic (Cardiac disorders) | 2 (3) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 2 (2)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Proteus infection (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cyst infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Retinal artery occlusion (Eye disorders) | 2 (2) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Rhinovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Varicella (Infections and infestations) | 2 (2) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular stent stenosis (General disorders) | 2 (3) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Venous stenosis (Vascular disorders) | 1 (3) | 1 (5)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorexia nervosa (Psychiatric disorders) | 0 (0) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 0 (0) | 1 (2)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous graft site abscess (Infections and infestations) | 1 (1) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
B-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (2) | 0 (0)
Benign neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Bone abscess (Infections and infestations) | 1 (1) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Boutonneuse fever (Infections and infestations) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burn infection (Infections and infestations) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Candida pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma in situ of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac discomfort (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0)
Catheter site abscess (Infections and infestations) | 1 (1) | 0 (0)
Catheter site oedema (General disorders) | 1 (1) | 0 (0)
Catheter site thrombosis (General disorders) | 0 (0) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral circulatory failure (Nervous system disorders) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Delayed graft function (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Device expulsion (Product Issues) | 0 (0) | 1 (1)
Device kink (Product Issues) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic microangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Discoloured vomit (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Douglas' abscess (Infections and infestations) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Endocarditis noninfective (Cardiac disorders) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia peritonitis (Infections and infestations) | 1 (1) | 0 (0)
External ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric mucosa erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal erosion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 0 (0) | 1 (1)
Graft loss (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic necrotic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic echinococciasis (Infections and infestations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
High turnover osteopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Implantation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1)
Infective aneurysm (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 1 (1) | 0 (0)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Keratorhexis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Listeraemia (Infections and infestations) | 0 (0) | 1 (1)
Listeria sepsis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Loss of personal independence in daily activities (Social circumstances) | 1 (1) | 0 (0)
Lumbar hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Measles (Infections and infestations) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mesenteric abscess (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mitral valve calcification (Cardiac disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Non-immune heparin associated thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ophthalmoplegia (Eye disorders) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (2)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Pachymeningitis (Nervous system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis infective (Infections and infestations) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vein occlusion (Vascular disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postictal state (Nervous system disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Protein C deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal artery thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst ruptured (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal transplant failure (Immune system disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus test positive (Investigations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal infection (Infections and infestations) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salmonella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Seizure cluster (Nervous system disorders) | 1 (1) | 0 (0)
Septic embolus (Infections and infestations) | 1 (1) | 0 (0)
Septic encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Serositis (General disorders) | 1 (1) | 0 (0)
Shigella infection (Infections and infestations) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt infection (Infections and infestations) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin weeping (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Streptococcal endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subendocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0)
Sympathetic ophthalmia (Eye disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Testicular infarction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Tolosa-Hunt syndrome (Eye disorders) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Ulcer (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Ulcerative gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureteric cancer regional (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vascular access site swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Vestibulitis (Infections and infestations) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=1482) | rhEPO (N=1474)
Hypertension (Vascular disorders) | 235 (366) | 232 (356)
Diarrhoea (Gastrointestinal disorders) | 161 (225) | 176 (228)
Headache (Nervous system disorders) | 115 (176) | 139 (216)
Dialysis hypotension (Vascular disorders) | 135 (254) | 105 (206)
Nasopharyngitis (Infections and infestations) | 113 (188) | 104 (188)
Arthralgia (Musculoskeletal and connective tissue disorders) | 101 (120) | 111 (138)
Hypotension (Vascular disorders) | 115 (140) | 92 (130)
Cough (Respiratory, thoracic and mediastinal disorders) | 101 (128) | 101 (133)
Upper respiratory tract infection (Infections and infestations) | 99 (144) | 92 (125)
Bronchitis (Infections and infestations) | 87 (116) | 97 (124)
Nausea (Gastrointestinal disorders) | 83 (95) | 84 (106)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 85 (105) | 76 (99)
Vomiting (Gastrointestinal disorders) | 83 (103) | 76 (98)
Fall (Injury, poisoning and procedural complications) | 73 (96) | 84 (119)
Back pain (Musculoskeletal and connective tissue disorders) | 64 (87) | 88 (103)
Urinary tract infection (Infections and infestations) | 73 (99) | 79 (97)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 61 (90) | 89 (121)
Hyperkalaemia (Metabolism and nutrition disorders) | 76 (92) | 62 (72)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 58 (67) | 74 (88)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT02879305/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT02879305/SAP_001.pdf